CLINICAL TRIAL: NCT05796726
Title: Retrospective Chart Review and Historical Comparison of Capmatinib vs. Standard of Care for German Adult Patients With Locally Advanced or Metastatic NSCLC Harboring METex14 Mutations
Brief Title: Retrospective Chart Review and Historical Comparison of Capmatinib vs. Standard of Care for German Adult Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC) Harboring METex14 Mutations
Acronym: RECAP
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CINC280ADE01
Record Dates: First submitted 2023-03-22; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Locally Advanced or Metastatic Non-Small Cell Lung Cancer Harboring METex14 Mutations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Capmatinib Patients: Patients who received first- or second-line treatment with capmatinib in Study GEOMETRY mono-1
- Standard of Care Patients: Patients who received appropriate comparative therapy (ACT) defined by the German HTA agency G-BA or standard of care (SoC) practiced in German routine care

SUMMARY:
The objective of the study was to compare the therapeutic benefit of capmatinib versus appropriate comparative therapy (ACT) defined by the German HTA agency G-BA for its benefit assessment of capmatinib but also versus the standard of care (SoC) practiced in German routine care. Due to its design as an adjusted, patient-level comparison, the RECAP study addresses the evidence gap due to the single-arm nature of pivotal evidence for capmatinib.

For this purpose, data on patients treated with ACT resp. SoC in German routine care has been collected via a retrospective chart review. This data was then used as an external control for a non-randomized, patient-level adjusted comparison with data from the GEOMETRY mono-1 study of capmatinib (NCT02414139).

Due to the non-interventional nature of this study, the definition of endpoints as primary or secondary was omitted formally.

ELIGIBILITY:
Inclusion criteria

* NSCLC (any histology)

  * METex14 mutation
  * Epidermal Growth Factor Receptor (EGFR) wildtype
  * Anaplastic lymphoma kinase (ALK) rearrangement negative
* Stage IV or Stage IIIB without indication for local therapy
* First or second line of treatment
* Age ≥18 years Exclusion criteria
* Prior treatment with crizotinib, capmatinib, tepotinib or other MET inhibitors
* Carcinomatous meningitis
* Symptomatic brain metastases
* Eastern Cooperative Oncology Group Status (ECOG) >1
* Uncontrolled, clinically significant heart diseases
* Malignant disease other than NSCLC within the past 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to an average of approximately 18 months
  OS was defined as time from start of treatment to death due to any cause. Per the protocol and due to the non-interventional nature of this study, outcome measures were not formally ranked as primary or secondary.
Progression-free survival (PFS) | Up to an average of approximately 18 months
  PFS was defined as time from start of treatment to first documented disease progression or death due to any cause. Per the protocol and due to the non-interventional nature of this study, outcome measures were not formally ranked as primary or secondary.
Time to central nervous system (CNS) progression (CNSprog) | Up to an average of approximately 18 months
  For patients without brain metastases at start of treatment, CNSprog was defined as time from start of treatment to first radiologically documented brain metastases. Per the protocol and due to the non-interventional nature of this study, outcome measures were not formally ranked as primary or secondary.
Overall response rate (ORR) | Up to an average of approximately 18 months
  For external control patients, ORR was defined as proportion of patients with a radiologically documented decrease in sum of tumor lesions (primary tumor and metastases). Decrease in sum of tumor lesions included complete cessation of any radiologically detectable tumor lesions.
  For GEOMETRY mono-1 patients, ORR was defined as proportion of patients with a best overall response as complete response (CR) or partial response (PR). CR and PR were assessed per RECIST 1.1 by BIRC. Per the protocol and due to the non-interventional nature of this study, outcome measures were not formally ranked as primary or secondary.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- Germany (10):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Giessen
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Würzburg